CLINICAL TRIAL: NCT05544604
Title: Effect of Motor Cortex Versus Insula Cortical Targets Stimulation Using Concentric Electrode Transcranial Direct Current Stimulation on Chronic Post-mastectomy Pain; a Randomized Sham Controlled Study
Brief Title: Motor Cortex Versus Insula Stimulation Using Transcranial Current Stimulation on Chronic Post-mastectomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Egypt Cancer Institute (Other)
Collaborators: Assiut University (Other)
Responsible Party: Principal Investigator, Mohannad Ahmed Mohamed, Principal Investigator, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 453
Record Dates: First submitted 2020-03-29; First posted 2022-09-16 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Post-Mastectomy Chronic Pain Syndrome
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: twenty patients will be randomly allocated into one of the study designed groups using serially numbered opaque closed envelopes. Each patient will be placed in the appropriate group after opening the corresponding sealed envelope. The patient will receive one of the following interventions either:
  * active tDCS (2 mA) targeting the primary motor cortex of the contralateral side of the pain for 20 minute duration for five sessions in five consecutive days (one session /day),
  * sham tDCS over the primary motor cortex in the same stimulation parameters will be used but the device will be turned off without patient knowledge after 30 seconds ,
  * active tDCS (2mA) targeting the insula of the contralateral side of the pain for 20 minute duration for five sessions in five consecutive days (one session /day),
  * sham tDCS over the insula in the same stimulation parameters will be used but the device will be turned off without patient knowledge after 30 seconds.
Who Masked: Participant, Outcomes Assessor
Masking Description: serially numbered opaque closed envelopes. Each patient will be placed in the appropriate group after opening the corresponding sealed envelope
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1: active primary motor cortex stimulation (Active Comparator): active tDCS (2 mA) targeting the primary motor cortex of the contralateral side of the pain for 20 minute duration for five sessions in five consecutive days (one session /day)
  Interventions: Device: Transcranial direct current stimulation
- group 2 : sham primary motor cortex stimulation (Sham Comparator): sham tDCS over the primary motor cortex in the same stimulation parameters will be used but the device will be turned off without patient knowledge after 30 seconds.
  Interventions: Device: Transcranial direct current stimulation
- group 3 : active insula stimulation (Active Comparator): active tDCS (2 mA) targeting the insula of the contralateral side of the pain for 20 minute duration for five sessions in five consecutive days (one session /day)
  Interventions: Device: Transcranial direct current stimulation
- group 4 : sham insula stimulation (Sham Comparator): sham tDCS over the insula in the same stimulation parameters will be used but the device will be turned off without patient knowledge after 30 seconds.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — tDCS will be delivered with current strength of 2 mA for 20 min . Current will be applied through two concentric electrodes target electrode; return electrode. First we will fill the electrode cage with an electroconductive gel, and then position the electrodes, with the target electrode over the FDI hotspot, and finally we fasten the electrodes with a tubular net-shaped elastic bandage in mesh tissue, making sure that it will not push the electrode forward or backward. This procedure will aim at reducing contact impedance and at creating a uniform adherence between the whole surface of the electrodes and the scalp, avoiding uneven distribution of the current (Fertonani, 2015). We will position the central electrode (anode) according to the study group over C3 or C4 , the stimulating electrode will be placed on the scalp at T7 or T8 for the insular cortex per the 10-20 (EEG) system.

SUMMARY:
This study is designed to evaluate the effect of two concentric electrode transcranial direct current stimulation over the primary motor cortex versus insular cortical targets in post mastectomy neuropathic pain.

DETAILED DESCRIPTION:
eighty patients within age group 18-65 years old with post mastectomy neuropathic pain that are resistant to medical treatment in the form of tramadol hydrochloride 100 mg twice daily, pregabalin 75 mg twice daily and Amitriptyline 25 mg once daily for at least two months or associated with significant adverse effect from medication will be involved in this study.

twenty patients will be randomly allocated into one of the study designed groups using serially numbered opaque closed envelopes. Each patient will be placed in the appropriate group after opening the corresponding sealed envelope. The patient will receive one of the following interventions either:

* active tDCS (2 mA) targeting the primary motor cortex of the contralateral side of the pain for 20 minute duration for five sessions in five consecutive days (one session /day),
* sham tDCS over the primary motor cortex in the same stimulation parameters will be used but the device will be turned off without patient knowledge after 30 seconds ,
* active tDCS (2mA) targeting the insula of the contralateral side of the pain for 20 minute duration for five sessions in five consecutive days (one session /day),
* sham tDCS over the insula in the same stimulation parameters will be used but the device will be turned off without patient knowledge after 30 seconds.

ELIGIBILITY:
Inclusion Criteria:

* eighty patients within age group 18-65 years old with post mastectomy neuropathic pain that are resistant to medical treatment in the form of tramadol hydrochloride 100 mg twice daily, pregabalin 75 mg twice daily and Amitriptyline 25 mg once daily for at least two months or associated with significant adverse effect from medication will be involved in this study.

Exclusion Criteria:

* We will exclude patients with intracranial metallic devices or with pacemakers or any other device. We also exclude those with extensive myocardial ischemia and those known to have epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
chronic postmastectomy pain relief | VAS monitoring after 5th session
  pain relief on the VAS after the 5th session
chronic postmastectomy pain relief | VAS monitoring after 15 days
  pain relief on the VAS after 15 days
chronic postmastectomy pain relief | VAS monitoring one month later
  pain relief on the VAS 1 month later

SECONDARY OUTCOMES:
VDS, LANSS and depression symptoms by HAM-D | VDS, LANSS and depression symptoms by HAM-D after 5th session
  VDS, LANSS and depression symptoms by HAM-D after the 5th session
VDS, LANSS and depression symptoms by HAM-D | VDS, LANSS and depression symptoms by HAM-D after 15 days
  VDS, LANSS and depression symptoms by HAM-D after 15 days
VDS, LANSS and depression symptoms by HAM-D | VDS, LANSS and depression symptoms by HAM-D after one month
  VDS, LANSS and depression symptoms by HAM-D 1 month later

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Mohamed Fares, Professor, Principal Investigator — South Egypt Cancer Institute
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No